CLINICAL TRIAL: NCT06003751
Title: A Phase 2a Study to Evaluate Safety and Tolerability After Single Administration of PER-001 Intravitreal Implant in Participants With Diabetic Retinopathy
Brief Title: A Study of PER-001 in Participants With Diabetic Retinopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Perfuse Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PER001-202
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Placebo sham
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 2 Cohort A (Experimental): Cohort A - Low Dose or Sham
  Interventions: Drug: PER-001 Intravitreal Implant - Low Dose; Drug: PER-001 Intravitreal Implant - Sham
- Phase 2 Cohort B (Experimental): Cohort B - High Dose or Sham
  Interventions: Drug: PER-001 Intravitreal Implant - High Dose; Drug: PER-001 Intravitreal Implant - Sham

INTERVENTIONS:
Drug: PER-001 Intravitreal Implant - Low Dose — PER-001 Low Dose Intravitreal Implant
  Arms: Phase 2 Cohort A
Drug: PER-001 Intravitreal Implant - High Dose — PER-001 High Dose Intravitreal Implant
  Arms: Phase 2 Cohort B
Drug: PER-001 Intravitreal Implant - Sham — PER-001 Intravitreal Sham

SUMMARY:
This is a Phase 2a, randomized, single-masked (participant), sham controlled clinical study.

DETAILED DESCRIPTION:
This clinical study is a randomized, single-masked (participant) study to further investigate the ocular and systemic safety and tolerability of the two dose levels of PER-001 Intravitreal Implants in participants with diabetic retinopathy. Participants who meet entry criteria will be randomized to receive either dose of PER-001 or sham control. A total of approximately 24 participants (12 in each Cohort, will be randomized).

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years of age at the time of signing the informed consent
* A negative pregnancy test for females of childbearing potential at Screening (serum) and Day 1 (urine).
* Best-corrected visual acuity (BCVA) of ≥ 60 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (Snellen equivalent of 20/63 or better) at Screening in potentially eligible eye(s) and prior to randomization at Day 1 in the study eye
* Moderately severe to severe non-proliferative diabetic retinopathy (NPDR) (diabetic retinopathy severity scale [DRSS] of 47 to 53) within the standard 7-field ETDRS.

Exclusion Criteria:

* Hemoglobin A1c >12%, or if HbA1c ≤12%, diabetes mellitus is uncontrolled in the opinion of the investigator
* Any condition which, in the opinion of the investigator, would preclude the participant's ability to comply with study requirements including completion of the study (including but not limited to diagnosis of dementia, Alzheimer's, and/or other neurological disease or physical incapacity)
* Females who are pregnant, nursing, or planning a pregnancy during the study
* Active cancer within past 12 months except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma or prostate cancer
* Uncontrolled blood pressure (defined as systolic >180 or diastolic >110 mmHg while the participant is sitting).
* Currently untreated diabetes mellitus or previously untreated participants who initiated oral anti-diabetic medication or insulin within 3 months prior to Day 1
* History of cerebrovascular accident or myocardial infarction within 6 months prior to Day 1
* Uncontrolled atrial fibrillation
* Systemic anti-VEGF treatment within 4 months prior to Day 1
* Any significant media opacity which precludes clinical evaluation and imaging of the retina
* Presence of centrally involved DME (within 500 μm of the foveal center) at Screening and Day 1
* Tractional retinal detachment, pre-retinal fibrosis, vitreomacular traction, or epiretinal membrane involving the fovea or disrupting the macular architecture
* Active rubeosis
* History of vitrectomy surgery or retinal detachment or macular hole (Stage 3 or 4)
* Uncomplicated cataract surgery within 3 months of Screening or yttrium-aluminum- garnet capsulotomy (YAG) within 4 weeks of Screening
* Aphakia or absence of posterior capsule
* Evidence of uncontrolled glaucoma (intraocular pressure must be < 25 mmHg) at Screening
* History of recurrent infectious or inflammatory ocular disease
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis (Note: mild blepharitis is permitted if stable)
* Any active uveitis and/or vitritis or history of idiopathic or autoimmune-associated uveitis
* History of herpetic ocular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Best-corrected Visual Acuity (BCVA) | End of Study(Week 24)
  Change in BCVA from Baseline at Week 24 using BETDRS or modified ETDRS chart (Charts 1, 2, and R as applicable) with standardized distance and lighting ill be used to calculate the LogMAR score
Intraocular Pressure (IOP) | End of Study(Week 24)
  IOP change from Baseline at Week 24 as measured by a calibrated Goldmann applanation tonometry.
Ocular Adverse events | End of Study(Week 24)
  Frequency, severity and timing of ocular adverse events reported during the study will have verbatim terms mapped to corresponding thesaurus terms from the Medical Dictionary for Regulatory Activities coding dictionary and reported in a table summary for each active and sham participants
Systemic Adverse events | End of Study(Week 24)
  Frequency, severity and timing of systemic adverse events reported during the study will have verbatim terms mapped to corresponding thesaurus terms from the Medical Dictionary for Regulatory Activities coding dictionary and reported in a table summary for each active and sham participants

CONTACTS AND LOCATIONS:
Locations (1):
- Perfuse Therapeutics, Inc, San Francisco, California, United States